CLINICAL TRIAL: NCT02566213
Title: Human Fine-motor-skills in Weightlessness: Comparison of a Laboratory and an Everyday-like Context
Acronym: FINESKILL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-084
Record Dates: First submitted 2015-07-28; First posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motor skills measurements (Other)
  Interventions: Other: Parabolic flight; Other: Motor skills measurements

INTERVENTIONS:
Other: Parabolic flight
Other: Motor skills measurements — * the kinematics measurements of the right hand with a motion analysis system;
  * the measurements of forces applied by the hand on the object to be grasped and moved with a 6 degree of freedom force sensor;
  * the measurement of position of the moved object with an inductive position encoder.

SUMMARY:
The human performance during weightlessness was tested in a multiplicity of laboratory experiments during parabolic flights and in space. It is therefore known that human fine motor skills as grasping are affected by the impact of changing gravity levels. However, because everyday life movements differ in several aspects from those done in an experimental lab situation, investigators do not know until know if this kind of movements is altered in the same extend.

Fine motor skills seem to depend on the context in which they are made. Thus, the performance in weightlessness during everyday life could substantially differ from the results given by previous laboratory studies.

This assumption will be tested in the present project, with subjects executing one and the same grasping movement in two different contexts, both in normal gravity conditions and in weightlessness. To that end, the investigators developed a new method which allows comparing the same grasping movements under different conditions.

DETAILED DESCRIPTION:
Investigations description Subjects sit at a table in front of a 15" computer screen, a centrally located joystick and a sliding lever on the right side. All devices are fixed to the table.

The subjects hand is fitted with six adhesive reflexive markers so that hand movements can be registered from above by two MX-F20 Vicon-Cameras, attached to a table-fixed metal frame. Lever forces are registered by an ATI Nano17 force transducers, lever fore-aft position by an inductive encoder, and eye position by an eye tracker (Tobii T60).

Subjects will perform two different tasks, one representing a typical laboratory (L), one an everyday-like task (E). In task L, a visual stimulus on the screen will prompt subjects to release the joystick, grasp the lever, move it forwards and back, and then return their hand to the joystick. In task E, subjects will use the joystick in a computer game ("spider chasing") and occasionally release the joystick, grasp the lever, move it forwards and back in order to collect a reward, and then return their hand to the joystick. In both tasks the visual stimuli are accompanied with acoustic signals. To hear these signals during the flight procedure, subjects are equipped with ear-phones, plugged into a laptop.

In one 20 second microgravity episode, task L will be performed five times or task E twice. The investigator starts each task with a click on the keyboard and it stops automatically after 20sec.

Control data will be registered from each subject for the same length of time during level flight at 1g.

During the whole test procedure the subject is not constraint in its natural behaviour except by an easy to open belt which fixes the subject to the chair. The subject can at any time end the experiment.

Equipment used For hand motion measurement and analysis we use a Vicon MX System, consisting of two MX20+ infrared high-speed cameras, each connected via cables with an MX Ultranet which processes the data. The Ultranet is connected with a network cable to a corresponding laptop (Dell).

Force is measured by a 6 degree of freedom force transducer which is part of an ATI DAQ F/T System, consisting of the force sensor Nano 17, a power supply box with booster and a 16-bit A/D converter (DAQ-Card, NI 6036E). It uses the PCMCIA bus of a second laptop (Fujitsu).

The position of the object to move is measured by an inductive position encoder (dc position encoder type 8740-5100 by burster).

The eye movement will be recorded by a standard USB-camera or a commercial eye-tracker (Tobii T60) when available.

All devices are commercially available and are used according their CE marking.

Experimental protocol Before flight subjects will be familiarised with the protocol. Two subjects will be studied during each flight. On ground, each subject gets 6 reflexive markers (6mm diameter) stuck on their right hand (4 on index, 2 on thumb, fixed with double sided adhesive tape).

The first subject takes a seat at the experimental set-up, the second one on an aircraft seat. The tested subject is then equipped with ear-phones plugged into a laptop. It helps to focus the attention on the tasks which are accompanied with acoustic signals. Recording devices are then adjusted to the subject by a standard calibration procedure, done by the test-operator. Before entering the first parabola the subject executes the same two grasping-tasks on level flight. After the first test parabola, during each 0g period it has to execute the grasping movements in one of each task - 4 parabolas task L with five episodes each, 10 parabolas task E with two episodes each. Entering the 0g phase the operator starts the test by a click on the keyboard, afterwards the tasks stop automatically. During 1g and 1,8g phases the test is interrupted. After the 15th parabola the subjects switch places and the second one starts with the tests during the 0g phases. On level flight back to the airport it executes the same two tasks again as control condition.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers (men or women),
* aged from 18 to 65,
* right handed,
* affiliated to a Social Security system and, for non-French resident, holding an European Health Insurance Card (EHIC)
* who accept to take part in the study,
* who have given their written stated consent,
* who have passed a medical examination similar to a standard aviation medical examination for private pilot aptitude. There will be no additional test performed for subject selection.

Exclusion Criteria:

* person who took part in a previous biomedical research protocol, of which exclusion period is not terminated,
* pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-10; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Gravity induced change in movement time (ms) | baseline
  Measured by 3D videocamera, it is the time between the beginning of the hand movement and the contact of the hand on the object
Gravity induced change in peak velocity of the hand (deg/sec) | baseline
  Measured by 3D videocamera
Gravity induced change in the maximum grip aperture of the hand (mm) | baseline
  Measured by 3D videocamera. It is the maximum distance between the first and the fifth digit before hand grasps the object
Gravity induced change in the initial force applied by the hand on the grasped object (newton) | baseline
  Force measured by a strain gauge

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France